CLINICAL TRIAL: NCT03160664
Title: Research on Optimization Program of Magnetic Seizure Therapy for Bipolar Mania Patients
Brief Title: Magnetic Seizure Therapy for Bipolar Mania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17411969900
Record Dates: First submitted 2017-05-14; First posted 2017-05-19 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder, Manic
Keywords: magnetic seizure therapy; electroconvulsive therapy; bipolar mania; cognition; randomized controlled trial
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnetic seizure therapy (Experimental): 8-10 treatment sessions of MST, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Device: Magpro X100 + Option; Other: treatment as usual (TAU)
- electroconvulsive therapy (Active Comparator): 8-10 treatment sessions of modified-ECT, three times per week in the first two weeks, two times per in the following two weeks.
  Interventions: Device: ThymatronSystem Ⅳ Electroconvulsive System; Other: treatment as usual (TAU)

INTERVENTIONS:
Device: Magpro X100 + Option — In addition to treatment as usual (TAU), participants were supposed to receive ten sessions of MST in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks.
  Other Names: magnetic seizure therapy
  Arms: magnetic seizure therapy
Device: ThymatronSystem Ⅳ Electroconvulsive System — In addition to treatment as usual (TAU), participants were supposed to receive ten sessions of modified ECT in four weeks, with three sessions per week in the first two weeks and two sessions per week in the following two weeks
  Other Names: electroconvulsive therapy
  Arms: electroconvulsive therapy
Other: treatment as usual (TAU) — Participants will engage in their inpatient treatment program as-usual.

SUMMARY:
This trial attempts to evaluate the treatment efficacy of magnetic seizure therapy (MST) and its safety for bipolar mania. Half of the participants will receive MST, while the other half will receive electroconvulsive therapy (ECT).

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) is likely to be an alternative options to electroconvulsive therapy (ECT).

Widespread stimulation of cortical and subcortical regions is inevitable for ECT since the substantial impedance of the scalp and skull shuts most of the electrical stimulus away from the brain. Nevertheless, magnetic pulses are capable to focus the stimulus to a specific area of the brain because they can pass the scalp and skull without resistance. In Addition, electric current will penetrate into deeper structures, while magnetic stimulus are only capable to reach a depth of a few centimeters. As a consequence, MST are able to generate focus stimuli on superficial regions of the cortex while ECT can't, which may give MST the capability to produce comparable therapeutic benefits with the absence of apparent cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of bipolar I disorder and currently in a manic episode;
2. convulsive therapy clinically indicated, such as severe psychomotor excitement or retardation, attempts of suicide, being highly aggressive, pharmacotherapy intolerance, and ineffectiveness of antipsychotics;
3. the Young Mania Rating Scale (YMRS) score ≥ 10;
4. informed consent in written form.

Exclusion Criteria:

1. primary diagnosis of other mental disorders;
2. severe physical diseases, such as stroke, heart failure, liver failure, neoplasm, and immune deficiency;
3. present with a laboratory abnormality that could impact on efficacy of treatments or safety of participants;
4. failure to respond to an adequate trial of ECT lifetime;
5. are pregnant or intend to get pregnant during the study;
6. Unremovable metal implants.
7. other conditions that investigators consider to be inappropriate to participate in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
changes in the Young Mania Rating Scale | At baseline, 4-week follow-up

SECONDARY OUTCOMES:
changes in the Repeatable Battery for the Assessment of Neuropsychological Status (rRBANS) | At baseline and 4-week follow-up
changes in the Montgomery Åsberg Depression Rating Scale (MADRS) | At baseline and 4-week follow-up
changes in the Clinical Global Impression Scale (CGI) | At baseline and 4-week follow-up
changes in the motor threshold (MT) | At baseline and 24 hours after the first treatment
  using single-pulse Transcranial Magnetic Stimulation (sTMS)
changes in brain gamma-aminobutyric acid （GABA）levels | At baseline, 24 hours after the first treatment, and at 4-week follow-up
  measured by Magnetic Resonance Spectroscopy (MRS)
changes in the resting state network | At baseline, 24 hours after the first treatment, and at 4-week follow-up
  measured by Magnetic Resonance Imaging (MRI)
changes in auditory evoked potentials (AEP) | At baseline and 24 hours after the first treatment
  measured by electroencephalogram (EEG)
changes in the Novel P300 | At baseline and 24 hours after the first treatment
  measured by electroencephalogram (EEG)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Sheng, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Sheng J, Yang F, Qiao Y, Wang W, Wen H, Yang Q, Chen X, Tang Y. Magnetic Seizure Therapy vs Modified Electroconvulsive Therapy in Patients With Bipolar Mania: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e247919. doi: 10.1001/jamanetworkopen.2024.7919. PMID 38683612